CLINICAL TRIAL: NCT02270437
Title: Safety and Efficacy of Cocktail Periarticular Injection for Pain Management in Simultaneous Bilateral Total Knee Arthroplasty- A Prospective, Randomized Trial
Brief Title: Safety and Efficacy of Cocktail Periarticular Injection in Simultaneous Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhihong Wu, Prof., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBX 726
Record Dates: First submitted 2014-08-02; First posted 2014-10-21 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Pain, Postoperative
Keywords: total knee arthroplasty; cocktail analgesia; morphine consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Fentanyl; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cocktail analgesia (Experimental): The local infiltration mixture of ropivacaine, fentanyl, adrenaline is used intra-articularly during operation. The patients in the cocktail analgesia group received an injection of 200mg ropivacaine, 100ug fentanyl, and 0.25mg adrenaline into knee collateral ligaments, posterior aspect of the capsule, quadriceps tendon, patellar tendon, fat pad, periosteum, and synovium, along with PCIA morphine postoperatively.
  Interventions: Drug: ropivacaine, fentanyl, adrenaline
- no cocktail injection (No Intervention): The patients in the no cocktail injection group received PCIA morphine postoperatively.

INTERVENTIONS:
Drug: ropivacaine, fentanyl, adrenaline — The patients in the cocktail analgesia group received an injection of 200mg ropivacaine, 100ug fentanyl, and 0.25mg adrenaline into knee collateral ligaments, posterior aspect of the capsule, quadriceps tendon, patellar tendon, fat pad, periosteum, and synovium, along with PCIA morphine postoperatively.
  Other Names: Naropin, AstraZeneca
  Arms: cocktail analgesia

SUMMARY:
We investigated the safety and efficacy of the bilateral periarticular cocktail injection at a reduced dosage in patients undergoing simultaneous bilateral total knee arthroplasty.

DETAILED DESCRIPTION:
It is hypothesized that intraoperative periarticular injection with cocktail analgesics can reduce postoperative parenteral narcotics use and improve patient satisfaction following total knee arthroplasty.

A prospective, randomized trial is conducted to testify the hypothesis above by recruiting patients who go through simultaneous bilateral TKA and observing their postoperative analgesic consumption, visual analog scores and functional recovery. Potential side-effects of the multimodal drugs is also under observation.

ELIGIBILITY:
Inclusion Criteria:

* patients with tricompartmental knee disease undergoing simultaneous bilateral TKA

Exclusion Criteria:

* diabetes mellitus
* neuromuscular deficit
* a known allergy to one of the drugs being injected
* a history of cardiac disease or arrhythmia requiring special monitoring

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the Morphine consumption and PCIA duration | 12 hours to 3 days after the surgery

SECONDARY OUTCOMES:
To evaluate the visual analog scale (VAS) in each group patients underwent total knee arthroplasty | 4 hours to 5 days after the surgery
Function recovery evaluation for patients received surgery | 1, 3 and 5 days after the surgery

OTHER OUTCOMES:
Testing of body temperature,routine blood examination | hospital admission and 1, 3, 5 days after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wu Zhihong, Prof, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China